CLINICAL TRIAL: NCT02734056
Title: Music During Labor Epidural Placement and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Bhavani Shankar Kodali, Anesthesiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001230
Record Dates: First submitted 2016-03-30; First posted 2016-04-12 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Satisfaction
MeSH Terms: conditions — Personal Satisfaction | interventions — Music Therapy

STUDY DESIGN:
Masking Description: No masking was possible.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music (Experimental): The intervention to be administered is music
  Interventions: Other: Music
- Control (Experimental): There is no intervention listed here because this is the control group, in which there will be no intervention.
  Interventions: Other: Control

INTERVENTIONS:
Other: Music — Listening to music that the patient likes
  Arms: Music
Other: Control — Control
  Arms: Control

SUMMARY:
Patient satisfaction is becoming increasingly important to hospital administrators as a metric for quality of patient care services because it is now being linked to reimbursements (Maher 2015). Patient satisfaction is a complex problem, and may be affected by a variety of factors. A recent study found that higher patient satisfaction was associated with patients who received music therapy during their hospital stay (Mandel 2014). Given that music may positively affect patient satisfaction, we are designing a study to examine the effects of patient-preferred music on patient satisfaction in women undergoing labor epidural placement.

DETAILED DESCRIPTION:
PROCEDURES STEP-BY-STEP

1. Once enrolled in the study, patient will be randomized to either:

   * The intervention group (music played on a portable speaker system), or
   * The control group (no music).
2. Prior to epidural placement, patients in both groups will be asked to answer one question about their music preference: "What is your favorite music? You can name an artist, genre, album, or any other identifier"

   • If patient preferred music is not available on the Pandora app, other apps will be searched (Spotify, Youtube, itunes Radio, etc.)
3. If patients are randomized to the intervention group, the investigator will create a station in the Pandora music app using the patient's preferred music. Volume will be initially set on low and portable speaker system placed within 3 feet of the patient (in order to ensure that she can hear the music). The music will be started and volume will then be adjusted to the patient's preference, avoiding music that is too loud but ensuring it is loud enough so the patient can hear it.
4. At that point, epidural placement will begin. Patients will receive an epidural in the normal fashion. Music will be continued throughout the duration of the epidural placement procedure, unless the patient requests that it be discontinued earlier.
5. If patients are randomized to the control group, no music will be played.
6. One hour after epidural placement, the patient will be asked to fill out the patient satisfaction survey to assess their satisfaction with the epidural placement. All patients from both the intervention and control group will be asked to complete the survey.
7. Data (see below) will be collected from the chart at time of enrollment and at time of study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women in labor

   • Healthy pregnant women in labor requesting epidural labor analgesia
2. >30 weeks gestation
3. Ages 18 - 45

Exclusion Criteria:

1. Any patient who refuses
2. Women with impaired decision-making capacity
3. Patients who are deaf or extremely hard of hearing (if patients wear a hearing aid and can hear with it, then patients are still eligible to be in the study)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Kodali, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Will publish in a medical journal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were consented prior to recruitment
Period: Overall Study
Arm/Group | Music | Control
Started | 50 | 50
Completed | 50 | 49
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Music | Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (6) | 32 (6) | 32 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 3 | 13
  White | 23 | 28 | 51
  More than one race | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Anxiety
Description: The questions will be scored and a composite score will be determined. The scale is the numeric rating score, from 0-10, where 0 represents no anxiety and 10 represents the worst anxiety. Unit of measure is score on a scale.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: NRS
Arm/Group | Music | Control
Number analyzed (Participants) | 50 | 49
NRS | 2.9 (3.3) | 1.4 (1.7)

ADVERSE EVENTS:
Time Frame: During the study period only
Description: No adverse events recorded
Arm/Group | Music | Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No